CLINICAL TRIAL: NCT04142918
Title: Diagnostic Markers of Neuropathic Odontalgia : Proof of Concept Study
Brief Title: Diagnostic Markers of Neuropathic Odontalgia
Acronym: DIAMOND-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AP-HP190545
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Oral Mucosa
Keywords: painful post-traumatic trigeminal neuropathy; neuropathic pain; neuropathic odontalgia; gingival biopsy
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Oral mucosa biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immunostaining — Immunostaining of oral mucosa/gingiva samples

SUMMARY:
The DIAMOND study aims to investigate the presence and diagnostic relevance of potential biomarkers of the blood-nerve barrier disruption as surrogate markers of painful post-traumatic trigeminal neuropathic pain in patients presenting with neuropathic odontalgia. The first part of the study explores the proof-of-concept and technical feasibility of intra-epithelial nerve fiber immunostaining in gingival/oral mucosa biopsies and the potential presence of these biomarkers in healthy patients (baseline condition).

DETAILED DESCRIPTION:
Painful Post-Traumatic Trigeminal Neuropathy (PPTTN) defines a neuropathic painful condition affecting the orofacial region, following local nerve trauma, usually secondary to dental treatments (tooth avulsion, root canal treatments….). It often presents as odontalgia of atypical presentation, unresponsive to conventional treatments. The diagnostic is often complex (and often is a diagnosis of elimination), leading to unnecessary iatrogenic dental treatments and insufficient pain relief.

This study aims to explore potential new markers of PPTTN, based on a translational approach following previous preclinical work that showed the importance of the disruption of the blood-nerve barrier in generating post-traumatic neuropathic pain. Several markers of such disruption have been highlighted (such as Claudin-5, Patched-1 and Frizzled-7) that could be specifically downregulated in neuropathic pain conditions (as compared to inflammatory neuritis conditions). As such, these markers could be interesting biomarkers of neuropathic pain. This study aims to explore the presence (and absence) of such markers in healthy vs neuropathic patients respectively.

The first part of the study investigates the technical feasibility of intra-epithelial nerve fiber staining in oral mucosa/gingiva specimens collected in healthy patients (undergoing routine oral surgery procedures) and the immunoreactivity/presence of such biomarkers in those specimens.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (over 18 years old) requiring an oral/dental surgical intervention that will generate gingival/mucosal tissue elimination (as part of the normal surgical procedure)

Exclusion Criteria:

* Patient with a diagnosed odontalgia
* Patient with Painful Post-Traumatic Trigeminal Neuropathy (PPTTN)
* Patient with unexplained pains or a neuropathic pain regardless of its location
* Patient under guardianship or trusteeship
* Patient who refuses to give his/her non-opposition to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring an oral/dental surgical intervention that will generate gingival/mucosal tissue elimination (as part of the normal surgical procedure)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Patched-1 Western Blot concentration | Baseline
  Patched-1 will be measured in oral mucosa/gingiva samples using Western Blot
Patched-1 immunohistochemistry concentration | Baseline
  Patched-1 will be measured in oral mucosa/gingiva samples using immunohistochemistry (IHC)
Patched-1 ELISA concentration | Baseline
  Patched-1 will be measured in oral mucosa/gingiva samples using ELISA
Frizzled-7 Western Blot concentration | Baseline
  Frizzled-7 will be measured in oral mucosa/gingiva samples using Western Blot
Frizzled-7 immunohistochemistry concentration | Baseline
  Frizzled-7 will be measured in oral mucosa/gingiva samples using immunohistochemistry (IHC)
Frizzled-7 ELISA concentration | Baseline
  Frizzled-7 will be measured in oral mucosa/gingiva samples using ELISA
Claudin-5 Western Blot concentration | Baseline
  Claudin-5 will be measured in oral mucosa/gingiva samples using Western Blot
Claudin-5 immunohistochemistry concentration | Baseline
  Claudin-5 will be measured in oral mucosa/gingiva samples using immunohistochemistry (IHC)
Claudin-5 ELISA concentration | Baseline
  Claudin-5 will be measured in oral mucosa/gingiva samples using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Nathan MOREAU, DDS, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bretonneau Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided